CLINICAL TRIAL: NCT01396395
Title: A Prospective, Multi-center, Random, Open-label Research on Nicorandil Treatment of Patients Diagnosed as CHD (Coronary Heart Disease) With Stable Angina
Brief Title: Research on Nicorandil Treatment of Patients Diagnosed as CHD (Coronary Heart Disease) With Stable Angina
Acronym: SIGMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR200101-501
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Stable Angina; Coronary Disease
Keywords: Nicorandil; Stable angina
MeSH Terms: conditions — Angina, Stable; Coronary Disease | interventions — Nicorandil

ARMS (2):
- Standard treatment plus nicorandil (Experimental): The subjects will receive nicorandil 5 milligram (mg ) tablet orally three times daily for a period of 12 weeks along with one of the standard antianginal therapies (such as aspirin, beta-blockers, lipid lowering statins and angiotensin-converting enzyme inhibitors [(ACEIs] as permitted by disease condition /as per standard local practices/prescribed per discretion of investigators).
  Interventions: Drug: Nicorandil; Drug: Standard Treatment
- Standard treatment (Other)
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Drug: Nicorandil — The subjects will receive Nicorandil 5 mg tablet orally three times daily for a period of 12 weeks along with the standard treatment.
  Arms: Standard treatment plus nicorandil
Drug: Standard Treatment — The subjects will receive one of the standard anti-anginal therapies which included but not limited to aspirin, ACEI, lipid lowering statins and beta blockers according to the recommendation of guidelines. If the subject's condition permitted, they should take all these medicines. However, the dose, route, frequency and duration were determined by investigators according to subject's specific condition.

SUMMARY:
This study of 402 cases of stable angina subjects who were diagnosed as Coronary Heart Disease (CHD) is a randomized, blank controlled, multi-center clinical study. Subjects who are taking standard treatment with stable symptoms will receive a 24-hour ambulatory electrocardiogram (ECG) (Holter) examination. They will be randomly divided into two groups. The nicorandil group will receive nicorandil 5 milligram (mg) (3 times a day = tid) on top of the standard treatment for 12 weeks, while the control group will stay on standard treatment. Nitrates and beta blockers need to be maintained on a stable dose. Other drugs that do not affect the primary endpoint may be adjusted per investigators decision.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be diagnosed as stable CHD, and must have at least one of these histories:

  1. A history of coronary revascularization Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Surgery at least 3 months ago
  2. Myocardial infarction
  3. More than 50 percent (%) stenosis detected by angiography
  4. Exercise Tolerance Testing (ETT) or Computed Tomography Angiography (CTA) showed more than 50% stenosis with typical angina symptoms
* Subjects must have at least 2 times of typical symptoms of myocardial ischemia occurred within a week Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Coronary syndrome or considering acute coronary syndrome (ACS)
* Left main coronary artery disease without revascularization
* Aortic stenosis
* Obstructive hypertrophic cardiomyopathy
* Subjects with hypertension systolic blood pressure (SBP) greater than (>) 170 millimeters of mercury (mmHg) or diastolic blood pressure (DBP) >100 mmHg) or hypotension (SBP less than [<] 90 mmHg or DBP<60 mmHg)
* Diagnosis as postural hypotension before
* Congestive heart failure (New York Heart Association [NYHA] class III - IV
* Ejection fraction (EF)<40% by Echocardiography
* Arrhythmias requiring active treatment
* Gastro-intestinal ulcer
* Concomitant medication such as Sulphonyl urea, PDE-5 inhibitor such as sildenafil, Trimetazidine for treatment of angina pectoris Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- For Locations in, Beijing, China

REFERENCES:
- [Derived] Jiang J, Li Y, Zhou Y, Li X, Li H, Tang B, Dai X, Ma T, Li L, Huo Y. Oral nicorandil reduces ischemic attacks in patients with stable angina: A prospective, multicenter, open-label, randomized, controlled study. Int J Cardiol. 2016 Dec 1;224:183-187. doi: 10.1016/j.ijcard.2016.08.305. Epub 2016 Aug 21. PMID 27657471

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 subjects randomized to standard+nicorandil group were included in standard group for safety analysis as they did not receive nicorandil. 1 subject randomized to standard group was included in standard+nicorandil group as nicorandil was received. Thus, safety set have 197 and 205 in Standard+nicorandil and standard group, respectively.
Groups:
- Standard Treatment Plus Nicorandil: The subjects received nicorandil 5 milligram (mg) tablet orally three times daily for a period of 12 weeks along with one of the standard antianginal therapies aspirin, beta-blockers, lipid lowering statins and angiotensin-converting enzyme inhibitors (ACEIs) as permitted by disease condition or as per standard local practices or prescribed per discretion of the investigators.
- Standard Treatment: The subjects received one of the standard antianginal therapies which included but not limited to aspirin, beta blockers, lipid lowering statins and ACEIs as permitted by disease condition or as per standard local practices or prescribed per discretion of investigators.
Period: Overall Study
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Started | 200 | 202
Safety Analysis Set | 197 (1 subject randomized to standard was included in standard+nicorandil as nicorandil was received.) | 205 (4 subjects randomized to standard+nicorandil were included in standard as no nicorandil was received)
Completed | 160 | 175
Not Completed | 40 | 27
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Protocol Violation | 3 | 1
Not completed — Adverse Event | 10 | 2
Not completed — Lost to Follow-up | 17 | 11
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized subjects who received at least one dose of study treatment.
Groups:
- Standard Treatment Plus Nicorandil: The subjects received nicorandil 5 mg tablet orally three times daily for a period of 12 weeks along with one of the standard antianginal therapies ( aspirin, beta-blockers, lipid lowering statins and angiotensin-converting enzyme inhibitors [ACEIs] as permitted by disease condition or as per standard local practices or prescribed per discretion of investigators.
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment | Total
Number analyzed (Participants) | 200 | 202 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (10.16) | 60.8 (9.94) | 61.1 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 74 | 132
  Male | 142 | 128 | 270

OUTCOME MEASURES:

1. Primary Outcome: Number of Myocardial Ischemia Attacks in 24 Hours
Description: Myocardial ischemia attack was evaluated by 24-hour Holter monitoring based on the following criteria: 0.08 seconds after the J point in electrocardiogram (ECG) or compared with baseline levels, ST-segment with horizontal or downward sloping down greater than or equal to (>=) 0.1 millivolts (mV), and lasted for >= 1 minute, and at least 1 minute of interval with another ischemic attack, as one array myocardial ischemia.
Time Frame: At Week 12
Population: FAS included all randomized subjects who received at least one dose of study treatment. N (number of subjects analyzed) signifies the number of subjects evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ischemic attacks per 24 hours
Groups:
- Standard Treatment Plus Nicorandil: The subjects received nicorandil 5 mg tablet orally three times daily for a period of 12 weeks along with one of the standard antianginal therapies (aspirin, beta-blockers, lipid lowering statins and angiotensin-converting enzyme inhibitors [ACEIs] as permitted by disease condition or as per standard local practices or prescribed per discretion of investigators).
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 141 | 150
ischemic attacks per 24 hours | 2.3 (8.46) | 3.8 (18.02)
Statistical Analysis 1: Comparison: Standard Treatment Plus Nicorandil vs Standard Treatment; Test type: Superiority or Other; p < 0.0001, poisson regression: Non-calibration mode; Ratio = 0.503, 95% CI 2-sided [0.435 to 0.581]
Statistical Analysis 2: Comparison: Standard Treatment Plus Nicorandil vs Standard Treatment; Test type: Superiority or Other; p = 0.0086, Poisson regression: Calibration model; Ratio = 0.503, 95% CI 2-sided [0.301 to 0.840]

2. Secondary Outcome: Change From Baseline in Total Myocardial Ischemic Burden at Week 12
Description: The total myocardial ischemic burden was defined as the product of the decrease, total array and total time of ST-segment in symptomatic and asymptomatic myocardial ischemia subjects within 24 hours.
Time Frame: Baseline, Week 12
Population: FAS included all randomized subjects who received at least one dose of study treatment. N (number of subjects analyzed) signifies the number of subjects evaluable for this outcome measure. Analysis was done only for subjects with myocardial ischemia attack.
Measure: Mean (Standard Deviation); unit: millimeter*minutes
Groups:
- Standard Treatment Plus Nicorandil: The subjects received nicorandil 5 mg tablet orally three times daily for a period of 12 weeks along with one of the standard antianginal therapies (aspirin, beta-blockers, lipid lowering statins and ACEIs as permitted by disease condition or as per standard local practices or prescribed per discretion of investigators).
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 133 | 146
millimeter*minutes | -38.63 (572.807) | 29.26 (404.070)

3. Secondary Outcome: Change From Baseline in Maximum ST-depression at Week 12
Description: The maximum ST- depression was evaluated from sum of all leads for all the subjects with myocardial ischemia attack. Absolute value of maximum ST-depression was used for calculation.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter
Groups:
- Standard Treatment Plus Nicorandil: The subjects received nicorandil 5 mg tablet orally three times daily for a period of 12 weeks along with one of the standard antianginal therapies ( aspirin, beta-blockers, lipid lowering statins and angiotensin-converting enzyme inhibitors [ACEIs] as permitted by disease condition or as per standard local practices or prescribed per discretion of investigators).
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 133 | 146
millimeter | 0.25 (3.598) | 0.36 (3.563)

4. Secondary Outcome: Change From Baseline in Longest Duration of ST Segment Depression at Week 12
Description: The maximum ST- depression was evaluated from sum of all leads for all the subjects with myocardial ischemia attack. The longest duration of ST segment depression of all leads for all the subjects with myocardial ischemia attack.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 133 | 146
seconds | -3.8 (37.75) | 3.4 (18.83)

5. Secondary Outcome: Percentage of Subjects Experienced Ischemic Heart Attack During the Six-minute Walk Test
Description: The percentage of subjects who experienced ischemic heart attack during the Six-minute walk test (6-MWT) were evaluated.The 6-MWT was the distance that a subject could walk in 6 minutes. Subjects were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. The 6-MWT was completed within 1-hour after wearing Holter.
Time Frame: At Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 135 | 147
percentage of subjects | 2.2 | 4.1

6. Secondary Outcome: Heart Rate Variability (HRV) Rate: Time Domain
Description: HRV is the degree of fluctuation in the length of the intervals between heart beats. All HRV parameters are calculated on 'normal-to-normal' (NN) inter-beat intervals (or NN intervals) caused by normal heart contractions. Standard deviation of all NN intervals (SDNN) and Standard deviation of the averages of NN intervals (SDANN) are the two time domain methods used to determine heart rate variability. Two variants of the SDNN, created by dividing the 24-hour monitoring period into 5-minute segments, are the SDNN index and the SDANN index. The SDNN index is the mean of all the 5-minute standard deviations of NN (normal RR) intervals during the 24-hour period, while the SDANN index is the standard deviation of all the 5-minute NN interval means.
Time Frame: At Week 12
Population: FAS included all randomized subjects who received at least one dose of study treatment. "n" signifies the number of subjects evaluable for each category in each group for this outcome measure, respectively.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 200 | 202
millisecond
  SDNN-24 hour (n=141, 149) | 126.1 (35.58) | 125.7 (33.25)
  SDANN index (n=141, 149) | 116.9 (37.44) | 116.7 (33.65)
  SDNN index (n=140, 147) | 47.6 (14.60) | 47.0 (14.99)

7. Secondary Outcome: Heart Rate Variability (HRV) Rate: Frequency Domain Power-24 Hour
Description: HRV is the degree of fluctuation in the length of the intervals between heart beats. All HRV parameters are calculated on 'normal-to-normal' (NN) inter-beat intervals (or NN intervals) caused by normal heart contractions. The HRV was evaluated based on frequency domain power-24 hours.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millisecond square (ms^2)
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 140 | 147
millisecond square (ms^2) | 2397.0 (1527.37) | 2328.6 (1458.31)

8. Secondary Outcome: Number of Arrhythmia Occurred Within 24 Hours
Description: The number of ventricular tachycardia and premature ventricular beats that occurred within 24 hours.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per 24 hours
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 141 | 150
beats per 24 hours
  Ventricular tachycardia | 0.8 (4.03) | 5.2 (40.67)
  Premature ventricular beat | 134.8 (457.59) | 569.1 (2538.17)

9. Secondary Outcome: ECG QT Dispersion
Description: The ECG QT dispersion was defined as the difference between the longest (QTmax) and the shortest (QTmin) QT intervals within a 12-lead ECG.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 74 | 69
milliseconds | 0.1298 (0.17240) | 0.1110 (0.15865)

10. Secondary Outcome: Number of Subjects Experienced Angina Attack
Time Frame: Baseline up to 12 Weeks
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 162 | 176
subjects | 48 | 70

11. Secondary Outcome: Frequency of Angina Attack
Description: The total number of times angina attacks occurred within a week (number of times/week)
Time Frame: At Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: angina attacks per week
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 45 | 70
angina attacks per week | 1 [1 to 2] | 2 [1 to 2]

12. Secondary Outcome: Number of Subjects Relieved From Angina Attack After the Consumption of Nitroglycerin
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 26 | 48
subjects | 20 | 43

13. Secondary Outcome: Number of Nitroglycerin Tablets Consumed in a Week
Time Frame: At Week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: tablets per week
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 19 | 43
tablets per week | 1 [1 to 4] | 2 [1 to 2]

14. Secondary Outcome: Walk Distance in Six Minute Walk (6-MWT) Test at Week 12
Description: The 6-MWT distance was the distance that a subject could walk in 6 minutes. Subjects were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. The 6-MWT was completed within 1-hour after wearing Holter.
Time Frame: At Week 12
Population: FAS included all randomized subjects who received at least one dose of study treatment. N (number of subjects analyzed) signifies number of subjects evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 152 | 164
meters | 452.1 (116.87) | 438.1 (107.42)

15. Secondary Outcome: Number of Subjects With Any Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Death, and AEs Leading to Discontinuation
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs were defined as the AEs that occurred between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study drug administration up to 30 days after the last dose of study drug administration (up to 16 weeks )
Population: Safety analysis population included all the subjects who received at least one dose of the study drug. 4 subjects randomized to standard+nicorandil group were included in standard group for safety analysis as they did not receive nicorandil. 1 subject randomized to standard group was included in standard+nicorandil group as nicorandil was received.
Measure: Number; unit: subjects
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Number analyzed (Participants) | 197 | 205
subjects
  TEAEs | 23 | 13
  SAEs | 9 | 7
  AEs Leading to Death | 1 | 1
  AEs Leading to Discontinuation | 16 | 0

16. Secondary Outcome: Number of Subjects Who Showed Compliance to Nicorandil
Description: Compliance percent (%) was calculated by using the formula: (actual total dose divided by planned total dose) multiplied by 100. If subject compliance was less than 80% or greater than 120%, then that subject was considered as non compliant. The compliance of subjects taking nicorandil was evaluated.
Time Frame: Baseline up to 12 Weeks
Population: as for outcome 15
Measure: Number; unit: subjects
Arm/Group | Standard Treatment Plus Nicorandil
Number analyzed (Participants) | 191
subjects | 181

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to 30 days after the last dose of study drug administration (up to 16 weeks ).
Arm/Group | Standard Treatment Plus Nicorandil | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 9/197 | 7/205
Other Adverse Events (participants affected / at risk) | 12/197 | 1/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment Plus Nicorandil (N=197) | Standard Treatment (N=205)
Sudden death (Cardiac disorders) | 1 | 0
Cardiac sudden death (Cardiac disorders) | 0 | 1
Angina (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Unstable angina (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Peripheral edema (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Diabetes (Metabolism and nutrition disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastroenteritis' (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Increased blood pressure (Investigations) | 1 | 0
Chronic renal failure (Renal and urinary disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment Plus Nicorandil (N=197) | Standard Treatment (N=205)
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 6 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Chest pain (Cardiac disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other